CLINICAL TRIAL: NCT01398449
Title: Is Elective Nodal Irradiation (ENI) Necessary For Patients With Thoracic Esophageal Squamous Cell Carcinoma Who Undergo Esophagectomy And With Pathological Stage Of T1-2,N+,M0 -- A Randomized Phase Ⅲ Trial
Brief Title: Is ENI Necessary For Patients With Thoracic Esophageal Cancer After Esophagectomy And With Pathological Stage Of T1-2,N+,M0
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Jiangsu Cancer Institute & Hospital (Other); Affiliated Hospital of Jiangsu University (Other); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Hospital (Other Government); Fujian Cancer Hospital (Other Government); Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); RenJi Hospital (Other)
Responsible Party: Xiao-Long Fu / Professor, Fudan University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011ESO_FU_02
Record Dates: First submitted 2011-07-13; First posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: thoracic esophageal squamous cell carcinoma; esophagectomy; elective nodal irradiation; adjuvant chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): After esophagectomy, patients in Arm B will receive adjuvant chemotherapy, followed by elective nodal irradiation (ENI)
  Interventions: Radiation: Elective nodal irradiation (ENI)
- A (Active Comparator): After esophagectomy, patients in Arm A will receive adjuvant chemotherapy only
  Interventions: Other: Adjuvant chemotherapy only

INTERVENTIONS:
Radiation: Elective nodal irradiation (ENI)
  Arms: B
Other: Adjuvant chemotherapy only
  Arms: A

SUMMARY:
Is elective nodal irradiation (ENI) necessary for patients with thoracic esophageal cancer after esophagectomy and with pathological stage of T1-2,N+,M0?

DETAILED DESCRIPTION:
Patient Population:

Thoracic esophageal squamous cell carcinoma after esophagectomy with at least 15 lymph nodes removed for adequate nodal staging.

R0 resection; T1-2, N+, M0.

Scheme:

After esophagectomy, patients are firstly stratified by numbers of lymph node metastasis (<3 or >=3). Then patients are randomized to 2 arms:

Arm A:

Adjuvant chemotherapy (4 cycles).

Arm B:

Adjuvant chemotherapy (4 cycles) + Elective Nodal Irradiation (bilateral supraclavicular fossa and mediastinum).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤70
2. ECOG performance status 0-1
3. Weight is not less than 90% of it before operation
4. Registration within 8 weeks after esophagectomy
5. Histologically proven primary thoracic esophageal squamous cell carcinoma
6. R0 resection and number of lymph nodes dissected ≥15 after esophagectomy
7. Stage T1-2N1-3M0 based pathological diagnosis
8. Chest and abdominal contrast enhanced CT within 6 weeks prior to registration(PET/CT scan is selective)
9. Without supraclavicular nodes and abdominal regions nodes existed after surgery
10. Without neo-adjuvant chemotherapy and radiotherapy
11. WBC≥ 4.0X109/L ,Absolute neutrophil count (ANC) ≥ 2.0X109/L
12. Platelets ≥ 100X109/L
13. Hemoglobin ≥ 90g/L(without blood transfusion)
14. AST (SGOT)/ALT (SGPT) ≤ 2.5 x upper limit of normal, Bilirubin ≤ 1.5 x upper limit of normal
15. Creatinine ≤ 1.5 x upper limit of normal
16. Sign study-specific informed consent prior to study entry

Exclusion Criteria:

1. Multiple primary esophageal tumors
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
3. Severe, active comorbidity, defined as follows:

   3.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months 3.2 Transmural myocardial infarction within the last 6 months 3.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration 3.4 Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration 3.5 Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
4. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
5. Prior systemic chemotherapy, prior radiation therapy or prior target drug therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 874 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival
  To evaluate elective nodal irradiation (ENI) is better for the overall survival of patients with thoracic esophageal cancer after esophagectomy who with pathological stage of T1-2, N positive, M0

SECONDARY OUTCOMES:
Locoregional control rate
Safety and Tolerability (incidence rate of adverse events)
  the incidence rate of adverse events, especially radiation-induced lung toxicity
Failure pattern
  To evaluate the rationality of ENI after esophagectomy by analyzing the therapeutic failure patterns especially by comparing the in-field and out-of-field recurrences

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China